CLINICAL TRIAL: NCT02199275
Title: Impact of General Anesthesia on Enterocyte Damage
Brief Title: Effect of General Anesthesia on Enterocyte Damage
Acronym: GUT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Principal Investigator, Gael PITON, MCU-PH, Centre Hospitalier Universitaire de Besancon
Other Study IDs: P/2013/174
Record Dates: First submitted 2013-09-04; First posted 2014-07-24 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Non-urgent Surgery; General Anesthesia
Keywords: Non-urgent surgery; General anesthesia; Enterocyte damage; Intestinal fatty acid-binding protein

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Blood samples on venous puncture
Oversight: Data Monitoring Committee: Yes

SUMMARY:
During non urgent surgery, general anesthesia might induce enterocyte damage. I-FABP is a performant biomarker of enterocyte damage. We aimed to study whether patient ongoing general anesthesia for non-urgent surgery have an elevation of plasma I-FABP concentration.

DETAILED DESCRIPTION:
Inclusion criteria

* Indication of non-urgent surgery
* General anesthesia protocol using propofol and remifentanyl
* One half of the patients have a history of ischemic arteriopathy
* One half of the patients have no history of ischemic arteriopathy

Exclusion criteria

* Age < 18 years old
* Pregnant

Primary objective

Is there a significant elevation of I-FABP between the pre-anesthesic period and 11 minutes after induction of general anesthesia ?

Secondary objectives

1. Is I-FABP elevation higher among patients with history of patent arteriopathy ?
2. Is I-FABP elevation higher among patients presenting with hypotension during anesthesia ?

ELIGIBILITY:
Inclusion criteria

* Indication of non-urgent surgery
* General anesthesia protocol using propofol and remifentanyl
* One half of the patients have a history of ischemic arteriopathy
* One half of the patients have no history of ischemic arteriopathy

Exclusion criteria

* Age < 18 years old
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults requiring non-urgent surgery, in whom a protocol of general anesthesia using propofol and remifentanyl with monitoring of bispectral index is expected.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
I-FABP elevation after induction of general anesthesia | 11 minutes
  Primary measure of plasma I-FABP before induction of general anesthesia. Second measure of plasma I-FABP concentration 11 minutes after induction of general anesthesia using a protocol of propofol and remifentanyl with monitoring of bispectral index.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Besançon, Besançon, France